CLINICAL TRIAL: NCT06643455
Title: Mindfulness Intervention for Nutrition in the Digital Kitchen (MIND) Study: A Pilot and Feasibility Study
Brief Title: Mindfulness Intervention for Improving Nutrition in the Digital Kitchen Among Stage I-III Breast Cancer Survivors, MIND Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: Apex Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RG1124573; NCI-2024-06603 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 0020593 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2024-09-27; First posted 2024-10-16 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Anatomic Stage I Breast Cancer AJCC v8; Anatomic Stage II Breast Cancer AJCC v8; Anatomic Stage III Breast Cancer AJCC v8
MeSH Terms: interventions — Practice Guidelines as Topic; Standard of Care; Electronic Health Records

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (MIND program) (Experimental): Patients participate in the MIND program consisting of self-paced online education on nutrition, chef demo skills-building cooking, and mindfulness practice over 4 hours weekly for 6 weeks.
  Interventions: Behavioral: Behavioral Dietary Intervention; Other: Electronic Medical Record; Other: Questionnaire Administration
- Arm B (waitlist control) (Active Comparator): Patients participate in SOC for 6 weeks. Patients may optionally receive access to the MIND program following the initial 6-week study period.
  Interventions: Other: Best Practice; Other: Electronic Medical Record; Other: Questionnaire Administration

INTERVENTIONS:
Behavioral: Behavioral Dietary Intervention — Participate in the MIND program
  Arms: Arm A (MIND program)
Other: Best Practice — Participate in SOC
  Other Names: standard of care; standard therapy
  Arms: Arm B (waitlist control)
Other: Electronic Medical Record — Ancillary studies
  Other Names: Computer Based Patient Record; EMR; EMR (electronic medical record)
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This trial tests how well a remotely-delivered nutrition and culinary intervention works to improve diet quality among stage I-III breast cancer survivors. Despite the strong evidence demonstrating the benefits of healthy nutrition on improving cancer outcomes, most breast cancer survivors, do not meet the nutrition recommendations The use of technology in behavioral interventions is proving to be a cost-effective mode of delivering lifestyle education to promote behavior change. The Mindfulness Intervention for Nutrition in the Digital Kitchen (MIND) program is delivered through a learning management system on the Cook for Your Life platform (cookforyourlife.org). The Cook for Your Life platform is a cancer patient-facing interactive program offering free nutrition and healthy cooking information, recipes, and cooking videos that disseminate evidence-based information on nutrition and cancer survivorship. The MIND program may help improve diet quality and increase fruit and vegetable intake among stage I-III breast cancer survivors.

DETAILED DESCRIPTION:
OUTLINE: Patients are randomized to 1 of 2 arms.

ARM A (INTERVENTION): Patients participate in the MIND program consisting of self-paced online education on nutrition, chef demo skills-building cooking, and mindfulness practice over 4 hours weekly for 6 weeks.

ARM B (WAITLIST CONTROL): Patients participate in standard of care (SOC) for 6 weeks. Patients may optionally receive access to the MIND program following the initial 6-week study period.

After completion of study intervention, patients are followed up at 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older.
* Previous diagnosis of stage I-III breast cancer in the past 5 years at the time of enrollment.
* No evidence of current, recurrent or metastatic disease.
* At least 60 days post final chemotherapy, biologic therapy, or radiation therapy and/or surgery. The following which are allowed: HER2-targeted therapies, CDK4/6 inhibitor (abemaciclib or ribociclib), endocrine therapy (aromatase inhibitors, ovarian suppression therapy, and tamoxifen), PARP inhibitors (olaparib), and bisphosphonates.
* Access to phone for study contacts.
* Access to smartphone, tablet, or computer and internet to attend online program.
* Willing and able to complete all study activities after randomization, including completing surveys online, at-home, or over the telephone.
* Able to understand and willing to sign written informed electronic (e) consent in English
* Eastern Cooperative Oncology Group (ECOG) status of 0-2.
* Participants must consume < 5 servings of fruits and vegetables per day as assessed by a brief questionnaire.
* At the time of enrollment, women must not be pregnant or lactating or planning to become pregnant in the next 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-05-16 (Actual); Primary Completion 2026-01-14 (Estimated); Study Completion 2026-01-14 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Accrued (Feasibility) | Up to 12 months
  Accrual of participants will be measured from date of initiating recruitment until last date of participant enrollment. Accrual will be considered feasible if enrollment goals (n=100 participants enrolled) is achieved in one year from initiation of recruitment.
Engagement (Feasibility) | Up to 12 weeks
  Will be considered feasible with if ≥ 70% of participants completing ≥ 70% of modules and attending ≥ 70% of live question and answer sessions. Baseline and demographics variables will be summarized by descriptive statistics. Binary proportions can be estimated to within 15% with 95% confidence intervals.
Retention (Feasibility) | Up to 12 weeks
  Will be considered feasible with if ≥ 70% of participants complete the week 6 food frequency questionnaire. Baseline and demographics variables will be summarized by descriptive statistics. Binary proportions can be estimated to within 15% with 95% confidence intervals.
Acceptability of Mindfulness Intervention for Nutrition in the Digital Kitchen (MIND) program | Up to 12 weeks
  Will be considered feasible with if ≥ 70% of participants state that the MIND program was acceptable, appropriate, and feasible. Baseline and demographics variables will be summarized by descriptive statistics. Binary proportions can be estimated to within 15% with 95% confidence intervals.

SECONDARY OUTCOMES:
Change in Diet Quality (Healthy Eating Index-2015) Score | Baseline to 6 weeks (intervention arm) or to week 12 (waitlist control arm)
  Participant diet quality will be assessed using the Food Frequency Questionnaire (FFQ). The FFQ provides the data that allows for calculating the Healthy Eating Index (HEI)-2015. The range of scores for the HEI-2015 is 0-100. A higher score is considered better and represents meeting more of the recommended dietary guidelines. Binary proportions will be compared between arms using a chi-squared test with the continuity correction. For continuous outcomes, between group comparisons will be made using linear regression methods and adjusting for baseline values.
Daily servings of fruit and vegetables | Baseline to 6 weeks (intervention arm) or to week 12 (waitlist control arm)
  Will be assessed using the FFQ. Binary proportions will be compared between arms using a chi-squared test with the continuity correction. For continuous outcomes, between group comparisons will be made using linear regression methods and adjusting for baseline values.
Frequency of cooking at home | Baseline to 6 weeks (intervention arm) or to week 12 (waitlist control arm)
  Will be self-reported by patient. Binary proportions will be compared between arms using a chi-squared test with the continuity correction. For continuous outcomes, between group comparisons will be made using linear regression methods and adjusting for baseline values.
Anxiety | Baseline to 6 weeks (intervention arm) or to week 12 (waitlist control arm)
  Will be measured using the Patient-Reported Outcomes Measurement Information System (PROMIS) Anxiety Short Form. Binary proportions will be compared between arms using a chi-squared test with the continuity correction. For continuous outcomes, between group comparisons will be made using linear regression methods and adjusting for baseline values.
Depression | Baseline to 6 weeks (intervention arm) or to week 12 (waitlist control arm)
  Will be measured using the PROMIS Depression Short Form. Binary proportions will be compared between arms using a chi-squared test with the continuity correction. For continuous outcomes, between group comparisons will be made using linear regression methods and adjusting for baseline values.
Cognitive function | Baseline to 6 weeks (intervention arm) or to week 12 (waitlist control arm)
  Will be measured using the PROMIS Cognitive Function Short Form. Binary proportions will be compared between arms using a chi-squared test with the continuity correction. For continuous outcomes, between group comparisons will be made using linear regression methods and adjusting for baseline values.
Sleep disturbance | Baseline to 6 weeks (intervention arm) or to week 12 (waitlist control arm)
  Will be measured using the PROMIS Sleep Impairment Short Form. Binary proportions will be compared between arms using a chi-squared test with the continuity correction. For continuous outcomes, between group comparisons will be made using linear regression methods and adjusting for baseline values.
Pain interference | Baseline to 6 weeks (intervention arm) or to week 12 (waitlist control arm)
  Will be measured using the PROMIS Pain Interference Short Form. Binary proportions will be compared between arms using a chi-squared test with the continuity correction. For continuous outcomes, between group comparisons will be made using linear regression methods and adjusting for baseline values.

CONTACTS AND LOCATIONS:
Overall Officials: Heather Greenlee, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No